CLINICAL TRIAL: NCT03286959
Title: Effect of Different Liners on Pulpal Outcome and Survival of Composite Restorations After Partial Caries Removal: A Randomized Controlled Study.
Brief Title: Effect of Liners on Pulpal Outcome and Restoration Survival After Partial Caries Excavation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, Principal, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shreyasingh
Record Dates: First submitted 2017-09-08; First posted 2017-09-19 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Reversible Pulpitis
MeSH Terms: interventions — Polymerase Chain Reaction; Calcium Hydroxide; Dycal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PCR WITH CALCIUM HYDROXIDE (Active Comparator): PCR WITH CALCIUM HYDROXIDE : A layer of dycal (dentsply) was placed adjacent to pulpal or axial wall after mixing as per manufacturer recommendations followed by etching and restoration with composite using incremental technique.
  Interventions: Procedure: PCR with calcium hydroxide
- PCR WITH RMGIC (Active Comparator): PCR WITH RMGIC: A layer of resin modified liner ( GC Fuji II ) was placed adjacent to pulpal or axial wall and light cured for 40 sec. afterwards the cavity was restored with composite as in other groups.
  Interventions: Procedure: PCR with RMGIC
- PCR WITH DIRECT COMPOSITE (Active Comparator): PCR WITH DIRECT COMPOSITE: After partial caries excavation , etching and bonding was done directly without using any liner and cavity was restored with composite as in other groups
  Interventions: Procedure: PCR with direct composite

INTERVENTIONS:
Procedure: PCR with calcium hydroxide
  Other Names: indirect pulp capping with dycal
  Arms: PCR WITH CALCIUM HYDROXIDE
Procedure: PCR with RMGIC
  Other Names: indirect pulp capping with RMGIC
  Arms: PCR WITH RMGIC
Procedure: PCR with direct composite
  Other Names: indirect pulp capping with adhesive restorations
  Arms: PCR WITH DIRECT COMPOSITE

SUMMARY:
Aim of the study was to determine the effectiveness of cavity liners regarding survival of restoration beneath composite restoration after partial caries removal in permanent teeth with deep caries and to evaluate and compare the pulp vitality outcome both clinically and radiologically with and without liners.

Study was conducted in Post Graduate Institute of Dental Sciences, Rohtak in department of Conservative Dentistry & Endodontics. Mature permanent mandibular molars with deep dentinal caries and without any signs of irreversible pulpitis were included in the study. After partial excavation of caries, patients were randomly allocated into three groups- RMGIC, CH and DIRECT COMPOSITE group and were restored according to standard protocol.

DETAILED DESCRIPTION:
AIM AND OBJECTIVES The present study aims to

1. Evaluate the success of partial caries excavation in mandibular molar teeth.
2. Evaluate and compare the clinical and radiographic success with RMGIC, calcium hydroxide and without liners after partial caries excavation.
3. Evaluate and compare the effect of liners on restoration survival after partial caries excavation.

MATERIALS AND METHODS Study subjects were recruited from OPD of Department of conservative dentistry and endodontics, PGIDS, Rohtak.

METHODOLOGY Prior to treatment, a thorough clinical and radiological examination was carried out and a thorough history was taken.

Clinical procedure:

Mature mandibular permanent molars exhibiting deep caries involving more than half or two thirds of dentin were chosen for the study.

The teeth were evaluated by periapical radiographs, periodontal probing, percussion test, and vitality assessment with thermal test and electric pulp test; teeth determined to have reversible pulpitis were included and with irreversible pulpitis were excluded.

All periapical radiographs were exposed by using constant kVP, mA, and exposure time (70 KVP, 8 mA, and 0.8 sec.) with a Rinn paralleling device.

After administration of local anesthesia, rubber dam isolation of the involved tooth was done and tooth was swabbed with betadiene. Carious tissue from lateral walls and dentino enamel junction was removed completely while a layer of soft carious dentin was left adjacent to pulpal or axial wall followed by cleaning with distilled water and drying with sterile filter paper. Then the teeth were randomised into three groups using a computer generated sheet.

GROUP I CH GROUP- The pulpal or axial wall was lined by a layer of dycal as per manufacturer directions and restored with composite restoration using incremental technique.

GROUP II RMGIC GROUP - A layer of resin modified GIC was placed adjacent to pulpal or axial wall and tooth restored as above.

GROUP III DIRECT COMPOSITE GROUP- Tooth was restored with composite restorations as above without placing any liner.

FOLLOW UP- The patients were recalled periodically at 1 month, 3 months, 6 months and 12 months after the procedure for clinical (post operative sensitivity, pain, tenderness, vitality) and radiographic (widening of periodontal ligament space and periapical radiolucency) evaluation. Also, the restoration survival was assessed using modified Hickel criteria where marginal staining, marginal adaptation, fractures and retention, secondary caries and post operative sensitivity were evaluated.

CRITERIA FOR SUCCESSFUL PULPAL OUTCOME A positive vitality test. No pain on percussion. No widening of periodontal ligament on periapical radiograph. No clinical or radiographic signs and/or symptoms of irreversible pulpitis and pulp necrosis.

CRITERIA FOR FAILURE No response to pulp vitality test. Teeth exhibiting clinical or radiographic signs and/or symptoms of irreversible pulpitis and pulp necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to participate in the study.
* Mature permanent mandibular molars with deep dentinal caries involving more than half or two thirds of dentin.

Exclusion Criteria:

* Primary teeth.
* Teeth with irreversible pulpitis (spontaneous pain) or pulp necrosis, chronic periodontitis, cracked tooth, internal or external resorption, calcified canals, associated with sinus tract, and furcation or apical radiolucency.
* Immuno-compromised, diabetic, pregnant and hypertensive patients.
* Positive history of antibiotic and analgesic use.

Ages: 14 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Actual)
Dates: Start 2016-11-06 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Evaluate and compare the clinical and radiographic success with different liners after partial caries excavation | The patients were recalled periodically at 1 month, 3months, 6 months and 12 months after the procedure.
  CRITERIA FOR SUCCESSFUL OUTCOME The Presence of positive response to vitality tests, absence of tenderness or spontaneous pain will be considered as clinical signs of success while absence of any radiolucency in periapical or furcation region or root resorptions as radiographic signs of successful outcome.
  CRITERIA FOR FAILURE The presence of negative vitality tests, spontaneous pain, fistula, swelling, mobility will be considered as clinical signs of failure while presence of any radiolucency in furcation or periapical region, internal or external root resorption as radiographic signs of failure.
  Although the procedure of partial caries excavation will be considered fully successful only when it shows successful outcome both from maintaining pulpal vitality as per primary outcome measures and intact restoration as per secondary outcome measures described below.

SECONDARY OUTCOMES:
Evaluate and compare the effect of different liners on survival of composite restorations after partial caries excavation. | The patients were recalled periodically at 1 month, 3months, 6 months and 12 months after the procedure.
  Treatment outcome will be judged on the basis of clinical findings and photographs recorded at the the baseline and at follow up visits on the basis of FDI criteria as described by Hickel et al.
  Primary measurement variable will be restoration Retention/Fractures. But the secondary measurable variables will also be evaluated namely Marginal adaptation, Marginal staining, Postoperative sensitivity and Recurrence of caries. Scoring will range from 1( very good), 2(good, after correction very good), 3(sufficient/satisfactory, minor shortcomings), 4 (unsatisfactory, but repairable) to 5 ( poor, replacement necessary). Restorations rated 4 or 5 in one of the criteria will be classified as clinically unacceptable, excluded from further assessment and will be repaired or replaced

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh S, Mittal S, Tewari S. Effect of Different Liners on Pulpal Outcome after Partial Caries Removal: A Preliminary 12 Months Randomised Controlled Trial. Caries Res. 2019;53(5):547-554. doi: 10.1159/000499131. Epub 2019 May 16. PMID 31096259